CLINICAL TRIAL: NCT01145534
Title: Phase 1 Study for Testing Efficacy of Cissus Verticillata L Infusion in Controlling Glucose Concentration
Brief Title: Evaluation of Cissus Verticillata L. Infusion in Controlling Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Rosana Araújo Rosendo, Federal University of Paraiba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPB-0346
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2008-08

CONDITIONS: Diabetes
Keywords: diabetes,; medicinal plants,; glucose
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glibenclamide (Active Comparator): Patients used 5 mg glibenclamide daily for 60 days
  Interventions: Drug: glibenclamide
- Experimental (Experimental): Patients ingested the infusion of Cissus verticillata L. prepared as 1 g in 150 mL of hot water for 10 min. This was done daily for 60 days
  Interventions: Other: medicinal plant infusion

INTERVENTIONS:
Drug: glibenclamide — 5 mg as pills, taken daily during the morning for 60 days
  Other Names: Glibenclamida, Legrand GE
  Arms: Glibenclamide
Other: medicinal plant infusion — INfusion fo Cissus verticillata L., 1 g in 150 mL water, ingested daily for 60 days.
  Other Names: popular plant name: Insulina
  Arms: Experimental

SUMMARY:
The purpose of this study was to investigate whether the infusion of a medicinal plant (Cissus verticillata L.) would be effective in reducing glucose levels in blood and saliva of type 2 Diabetes patients.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is regarded as one of the most prevalent disease of the adult population. In many developing countries, this condition is regarded as major public health problem. Type 2 diabetes is a metabolic disorder characterized by high blood glucose related with a condition of insulin resistance and relative insulin deficiency. As Diabetes progresses, medications are necessary to control glucose levels.

The aim of this study was to investigate whether the infusion of a medicinal plant (Cissus verticillata L.) would be as effective as a regular drug (glibenclamide) in reducing glucose levels in blood and saliva of type 2 Diabetes patients. Several medicinal plants have been used as potential medication for controlling glucose levels in Diabetes patients. Few studies have explored this effect related to Cissus verticillata L.infusion, though it has been indicated by folk medicine of some Latin American countries.

ELIGIBILITY:
Inclusion Criteria:

* subjects of 30 up to 80 years of age
* positive diagnostic for type 2 diabetes mellitus (blood glucose level above 126 mg/dL)
* patients that signed the informed consent

Exclusion Criteria:

* patients with renal and hepatic disfunction,
* patients with cardiac problems or other systemic alterations (allergies, pulmonary and gastrointestinal problems)
* pregnant women

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
blood glucose | 60 days
  Blood glucose was measured using a Gluco Dr. Plus (AGM-3000) Blood Glucose Monitoring System.

SECONDARY OUTCOMES:
Salivary glucose level | 60 days
  The level of glucose in saliva was measured in laboratory after colleting non-stimulated saliva in test tubes.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio C Sampaio, PhD, Study Chair — Federal University fo Paraiba
Locations (1):
- Centro de Especialidades Odontologicas, Patos, Paraíba, Brazil

REFERENCES:
- See also: Official research group for studies related to medicinal plants — http://www.ccs.ufpb.br/gefao/